CLINICAL TRIAL: NCT02621112
Title: Efficacy of Intradermal Hepatitis B Vaccine in Renal Failure Patients
Brief Title: HBV Vaccine in Renal Failure Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UW 11-209
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intradermal HBVv with imiquimod (Experimental): Intradermal hepatitis B vaccination with topical imiquimod pretreatment. Subjects to receive intradermal 10mcg of recombinant hepatitis B vaccine at two separate sites (5mcg) with topical imiquimod ointment pretreatment 5 minutes before injection at 0, 1, 3, 6 months
  Interventions: Biological: Intradermal HBVv with imiquimod
- Intradermal HBVv with aqueous cream (Active Comparator): Intradermal hepatitis B vaccination with topical aqueous cream. Subjects to receive intradermal 10mcg of recombinant hepatitis B vaccine at two separate sites (5mcg) with topical aqueous cream pretreatment 5 minutes before injection at 0, 1, 3, 6 months
  Interventions: Biological: Intradermal HBVv with aqueous cream
- Intramuscular HBVv with aqueous cream (Active Comparator): Intramuscular hepatitis B vaccination with topical aqueous cream. Subjects to receive intramuscular 10mcg of recombinant hepatitis B vaccine at two separate sites (5mcg) with topical aqueous cream pretreatment 5 minutes before injection at 0, 1, 3, 6 months
  Interventions: Biological: Intramuscular HBVv with aqueous cream

INTERVENTIONS:
Biological: Intradermal HBVv with imiquimod — Intradermal hepatitis B vaccine with imiquimod pretreatment
  Arms: Intradermal HBVv with imiquimod
Biological: Intradermal HBVv with aqueous cream — Intradermal hepatitis B vaccine with aqueous cream pretreatment
  Arms: Intradermal HBVv with aqueous cream
Biological: Intramuscular HBVv with aqueous cream — Intramuscular hepatitis B vaccine with aqueous cream pretreatment
  Arms: Intramuscular HBVv with aqueous cream

SUMMARY:
Hepatitis B virus infection remains an important clinical issue among patients on renal replacement therapy. Seroconversion rate as defined by an anti-HBs Ab titer > 10 IU/L after intramuscular hepatitis B vaccination (HBVv) remains poor in this cohort. Factors associated with inadequate anti-HBs response include older age, diabetes mellitus, obesity and low hepatitis B vaccine dose. Various small-scale studies including multiple high dose intramuscular vaccination or multiple small dose intradermal vaccination were attempted with variable response. Recent study on dose sparing seasonal influenza vaccine delivered via a novel intradermal microneedle has demonstrated good immunogenic responses similar to full-dose intramuscular vaccination. Imiquimod, a synthetic TLR7 agonist useful for the treatment of DNA virus infection, has been shown to improve vaccine immunogenicity. The investigators therefore propose a prospective, randomized study to compare the safety and immunogenicity of intradermal hepatitis B vaccination with this novel device with intramuscular in patients on renal replacement therapy.

DETAILED DESCRIPTION:
The investigators aim to recruit at least 120 subjects on renal replacement therapy in this prospective double blind randomized controlled trial. All recruited subjects have to be HBsAg and anti-HBs negative before recruitment. Subjects were randomly assigned to three groups.

All patients received 4 doses of hepatitis B vaccine at 0,1,3 and 6 months: Group 1: to receive intradermal 10mcg of recombinant hepatitis B vaccine at two separate sites (5mcg) with topical imiquimod ointment pretreatment 5 minutes before injection. Group 2: to receive intradermal 10mcg of recombinant hepatitis B vaccine at two separate sites (5mcg) with topical placebo aqueous cream pretreatment 5 minutes before injection. Group 3: to receive intramuscular 10mcg (1mL) of recombinant hepatitis B vaccine at two separate sites (5mcg) with topical placebo aqueous cream pretreatment 5 minutes before injection.

Subjects will be advised not to wash the topical treatment for 8 hours after vaccination. Patients and investigators will be blinded to the type of topical treatment applied. Anti-HBs titre will be measured at baseline, before each vaccination, and at 12 and 18 months after the first dose of vaccination.

The primary end point is the seroprotection rate of the HBVv at 12 months after the first dose of vaccination. The secondary end points are the seroprotection rate of HBVv and the geometric mean titre (GMT) fold increase of the anti-HBs at 1, 3, 6, 12 (GMT only) and 18 months after the first dose of vaccination. Adverse reactions of the vaccine will also be assessed immediately and for 1 month after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Patients recruited have to be aged ≥ 21 years, with history of chronic renal failure and on renal replacement therapy (continuous ambulatory peritoneal dialysis or hemodialysis).
* All patients have to give written informed consent and will have up to 1 week period to decide.
* Subjects must be available to complete the study and comply with study procedures.
* Patients are willing to allow for serum samples to be stored beyond the study period, for potential additional future testing to better characterize immune response.
* All recruited subjects have to be HBsAg, anti-HBs and anti-HIV negative before recruitment.

Exclusion Criteria:

* Inability to comprehend and to follow all required study procedures
* History or any illness that might interfere with the results of the study or pose additional risk to the subjects due to participation in the study.
* Have a recent history (documented, confirmed or suspected) of a flu-like disease within a week of vaccination.
* Have a known allergy to components of the Study Vaccines.
* Have a positive urine or serum pregnancy test within 24 hours prior to vaccination, or women who are breastfeeding.
* Have an active neoplastic disease or a history of any hematologic malignancy.
* Have known chronic active hepatitis B and hepatitis C (HBsAg+ve and anti-HCV+ve).
* Have known active human immunodeficiency virus (HIV).
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in this study or expect to receive an experimental agent during this study.
* Unwilling to refuse participation in another clinical study through the end of this study.
* Axillary temperature ≥ 38°C or oral temperature ≥ 38.5°C within 3 days of intended study vaccination.
* Have a history of alcohol or drug abuse in the last 5 years.
* Have any condition that the investigator believes may interfere with successful completion of the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2016-01; Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Seroprotection rate to HBV | 12 months after first dose of hepatitis B vaccine
  percentage of recruited subjects with anti-HBs >10 mIU/mL

SECONDARY OUTCOMES:
Adverse reaction to hepatitis B vaccine | 1 month
Seroprotection rate to HBV | 1, 3, 6 and 18 months after first dose of hepatitis B vaccine
  percentage of recruited subjects with anti-HBs >10 mIU/mL
GMT fold increase of anti-HBs | 1, 3, 6, 12 and 18 months after first dose of hepatitis B vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Ivan FN Hung, MD FRCP, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Hung IF, Yap DY, Yip TP, Zhang RR, To KK, Chan KH, Tang SC, Lui SL, Levin Y, Kochba E, Lau JY, Yuen MF, Chan TM, Yuen KY. A Double-blind, Randomized Phase 2 Controlled Trial of Intradermal Hepatitis B Vaccination With a Topical Toll-like Receptor 7 Agonist Imiquimod, in Patients on Dialysis. Clin Infect Dis. 2021 Jul 15;73(2):e304-e311. doi: 10.1093/cid/ciaa804. PMID 32556176